CLINICAL TRIAL: NCT01493206
Title: A Prospective Single Arm Study of Intraoperative Radiotherapy for Locally Advanced or Recurrent Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMCC04/16
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Malignant Rectal Neoplasm; Recurrent Tumor
Keywords: intraoperative radiotherapy
MeSH Terms: conditions — Rectal Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intraoperative radiotherapy (Experimental)
  Interventions: Radiation: intraoperative radiotherapy

INTERVENTIONS:
Radiation: intraoperative radiotherapy — intraoperative radiotherapy

SUMMARY:
The hypothesis is that intraoperative radiotherapy for locally advanced or recurrent rectal cancer improve outcomes without causing significant side effects.

DETAILED DESCRIPTION:
Primary Outcome measures are 3-year locoregional control, progression-free and overall survival rates.

Secondary outcome measures are toxicities scores up to 3 months after surgery (acute) and greater than 3 months after surgery (late). Data collected at 3-6 month intervals for 30 months

ELIGIBILITY:
Inclusion Criteria:

* locally advanced or recurrent rectal cancer
* suitable for radical surgery but at high risk of positive resection margins,
* no evidence of metastasis,
* age greater than 18 years,
* histologically confirmed adenocarcinoma,
* ECOG performance status <2.
* Informed consent

Exclusion Criteria:

* unresectable pelvic disease
* distant metastasis
* significant co-morbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
clinical outcomes | 3-year
  locoregional control, progression-free and overall survival rates.

SECONDARY OUTCOMES:
toxicities | 3-6 monthly up to 30 months
  Toxicity score criteria defined by Intraoperative Radiation Therapy Working Group Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Sam Ngan, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia